CLINICAL TRIAL: NCT01368692
Title: Effect of Shoulder Retraction on Success Rate of Subclavian Vein Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-1103-124-357
Record Dates: First submitted 2011-05-22; First posted 2011-06-08 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Subclavian Vein Catheterization
Keywords: subclavian vein catheterization success rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- neutral shoulder (Active Comparator): neutral shoulder position during subclavian vein catheterization
  Interventions: Procedure: position of neutral shoulder
- shoulder retraction (Experimental): position of shoulder retraction during subclavian vein catheterization
  Interventions: Procedure: position of shoulder retraction

INTERVENTIONS:
Procedure: position of shoulder retraction — position of shoulder retraction by placing a saline bag between the scapula
  Arms: shoulder retraction
Procedure: position of neutral shoulder — neutral shoulder position during subclavian vein catheterization
  Arms: neutral shoulder

SUMMARY:
The purpose of this study is to determine whether the shoulder retraction by placing a saline bag between the scapula influences a success rate of subclavian vein catheterization.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing neurosurgery or thoracic surgery that requires the placement of subclavian venous catheterization

Exclusion Criteria:

* infection over the puncture site
* history of prior clavicular fracture
* anatomical anomaly of subclavian vein

Ages: 16 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
catheterization success rate | immediately after catheterization (an expected average of 1 hour)
  Subclavian vein catheterization will be performed after the induction of anesthesia and before the start of surgery.

SECONDARY OUTCOMES:
location of catheter tip | an expected average of one day after surgery
  Postoperative chest X-ray will be taken to check for the location of catheter tip immediately after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim HJ, Jung SH, Min J, Hong DM, Jeon Y, Bahk JH. Comparison of the neutral and retracted shoulder positions for infraclavicular subclavian venous catheterization: a randomized, non-inferiority trial. Br J Anaesth. 2013 Aug;111(2):191-6. doi: 10.1093/bja/aet026. Epub 2013 Mar 10. PMID 23479675